CLINICAL TRIAL: NCT01266928
Title: Does Vitamins C and E Supplementation of After Preterm Rupture of Membranes Prolong the Duration of Latency? A Prospective Randomized Controlled Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, M.D, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: gungorduk10
Record Dates: First submitted 2010-12-20; First posted 2010-12-24 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Preterm Premature Rupture of Membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitaminCE (Active Comparator): Eligible and consenting women were randomly assigned to capsules containing a combination of 1,000 mg vitamin C (ascorbic acid) and 400 international units of vitamin E (RRR alpha tocopherol acetate)
  Interventions: Drug: vitamine C and E
- no drug (No Intervention): no drug

INTERVENTIONS:
Drug: vitamine C and E — Eligible and consenting women were randomly assigned to capsules containing a combination of 1,000 mg vitamin C (ascorbic acid) and 400 international units of vitamin E (RRR alpha tocopherol acetate)
  Arms: vitaminCE

SUMMARY:
Preterm premature rupture of membranes (PPROM) is a complication affecting 3-4.5% of all pregnancies. PPROM is the main known cause of preterm delivery and is associated worldwide with increased rates of neonatal and maternal morbidity and mortality. Despite its frequency, very little is known about its pathophysiologic mechanisms. Mechanical strength is provided to fetal membranes by an extracellular collagen matrix. Types I, II, III and IV are the main collagen types in these membranes. Studies have shown that total collagen content is reduced in the amnion of women with preterm PROM.

Vitamin C is involved in the metabolism of collagen and has been proposed to play an important role in the maintenance of the integrity of the chorioamniotic membranes. Vitamin E may play a synergic role with vitamin C, increasing the antioxidant capacity against reactive oxygen. Woods et al hypothesized that an increase in dietary consumption or supplementation of vitamin C and E during pregnancy might reduce the risk of that portion of preterm PROM that may be mediated by oxidative injury to fetal membranes. Plessinger et al report that pretreatment of human amnion-chorion with vitamins C and E prevents hypochlorous acid-induced membrane damage.

Borna et al. reported a randomized, double-blind controlled study of vitamin C and E supplementation, in which women with preterm rupture of membranes and singleton gestations at 26 to 34 weeks were randomized to vitamin C and E supplementation or placebo. Supplementation with vitamin C and E were associated with longer latency before delivery. However, the sample size in this study was very small.

The aim of this study was to evaluate the effect of supplementation with vitamins C and E after preterm premature rupture of membranes. We hypothesised that supplementation vitamins C and E may be effective in decreasing oxidative stress and increasing the latency period.

ELIGIBILITY:
Inclusion Criteria:

Patients with a single nonanomalous fetus and PPROM at ≥ 24.0 and ≤ 34.0 weeks' gestation.

Exclusion Criteria:

fetus with anomalies, chorioamnionitis, experienced PPROM within 14 days of either amniocentesis or cervical cerclage placement, multiple gestation, obstetrical indication for immediate delivery, delivery within 24 h of admission intrauterine fetal death at the time of presentation.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
latency until delivery | 7 days
  The primary outcome was the latency until delivery

SECONDARY OUTCOMES:
postpartum endometritis rate, early onset neonatal sepsis rate, | days
  Other outcomes were the birth weight, mode of delivery, occurrence of clinical chorioamnionitis, postpartum endometritis, early onset neonatal sepsis, grade 3-4 intraventricular haemorrhage (IVH), stage 2-3 necrotizing enterocolitis (NEC), admission to intensive care unit (ICU), duration of stay in an intensive care unit and respiratory distress syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırkoy Women and Children Hospital, Istanbul, Bakırkoy, Turkey (Türkiye)